CLINICAL TRIAL: NCT06325592
Title: Association Between Surgical Timing and Route of Total Hysterectomy After Loop Electrosurgical Excision Procedure and Perioperative Risk in Patients With Cervical High-grade Squamous Intraepithelial Lesion
Brief Title: Association Between Surgical Timing and Route of Total Hysterectomy After LEEP and Perioperative Risk in Patients With Cervical HSIL
Status: Completed | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Dengfeng Wang, Director of the first ward of Gynecology Oncology Department, Sichuan Cancer Hospital and Research Institute
Other Study IDs: REHSIL2023V1.1
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: High-Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- group 1: patients underwent laparoscopic hysterectomy within 3 days after LEEP
  Interventions: Procedure: surgical timing and operation path
- group 2: patients underwent abdominal hysterectomy within 3 days after LEEP
  Interventions: Procedure: surgical timing and operation path
- group 3: patients underwent laparoscopic hysterectomy 4 weeks after LEEP
  Interventions: Procedure: surgical timing and operation path
- group 4: underwent abdominal hysterectomy 4 weeks after LEEP
  Interventions: Procedure: surgical timing and operation path
- control group: Patients who underwent laparoscopic hysterectomy (LH) due to benign gynecological diseases were included in the control group.

INTERVENTIONS:
Procedure: surgical timing and operation path — surgical timing; laparoscopic hysterectomy or abdominal hysterectomy
  Groups: group 1; group 2; group 3; group 4

SUMMARY:
This study aimed to analyze perioperative information in patients with high-grade squamous intraepithelial lesion (HSIL) undergoing total hysterectomy (TH), offering insights into optimal surgery timing, selecting the operation path, and enhancing surgical operation details.

ELIGIBILITY:
Inclusion Criteria:

* patients were confirmed with HSIL through pathology at our hospital or another tertiary facility, with additional confirmation via pathological consultation at our facility;
* LH or abdominal hysterectomy (AH) +/- bilateral fallopian tube or bilateral adnexectomy was performed after LEEP;
* the patient had no history of systemic malignancies.

Exclusion Criteria:

* severe medical and surgical complications;
* an extensive or subextensive hysterectomy was performed;
* surgical removal scope involving tissues (such as lymph nodes) or organs (such as the appendix) other than the uterus, ovaries, and fallopian tubes;
* fever symptoms within the last month;
* incidence of pelvic and abdominal infections, vaginitis, or similar conditions within the past month.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gynecological patient
Study Population: Data were collected from patients with HSIL who underwent TH at the Gynecological Oncology Center of Sichuan Cancer Hospital between January 1, 2016, and October 31, 2023. Patients who underwent laparoscopic hysterectomy (LH) +/- bilateral fallopian tubes or bilateral adnexectomy for benign gynecological diseases (such as uterine fibroids and adenomyosis) were included in the control group (excluding patients with recent invasive operations of the cervix and vagina).
Sampling Method: Non-Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative fever | Within 7 days of surgery
  Use a thermometer to measure your temperature
Postoperative therapeutic use of antibiotics | Within 7 days of surgery
  Postoperative therapeutic use of antibiotics

SECONDARY OUTCOMES:
Postoperative complications | Within 7 days of surgery
  Postoperative complications
Postoperative hospitalization days | Date of surgery to date of discharge
  Postoperative hospitalization days
Postoperative hemoglobin | Within 7 days of surgery
  Postoperative hemoglobin
Postoperative white blood cell count | Within 7 days of surgery
  Postoperative white blood cell count
Postoperative erythrocyte count | Within 7 days of surgery
  Postoperative erythrocyte count
Postoperative albumin number | Within 7 days of surgery
  Postoperative albumin number
Postoperative CRP value | Within 7 days of surgery
  Postoperative CRP value

CONTACTS AND LOCATIONS:
Overall Officials: Dengfeng Wang, Ph.D, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No